CLINICAL TRIAL: NCT02768220
Title: The Effect of Sodium-Glucose Cotransporter 2 Inhibitors on Advanced Glycation End Products
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Caroline Messer, MD, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2-AGE
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: SGLT-2 Inhibitors; Advanced Glycation End Products; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Linagliptin (Active Comparator): Eligible patients were randomized to receive linagliptin 5mg daily for 30 days.
  Interventions: Drug: empagliflozin
- Empagliflozin (Experimental): Eligible patients were randomized empagliflozin 25mg daily for 30 days.
  Interventions: Drug: linagliptin

INTERVENTIONS:
Drug: empagliflozin — Test to see how 30 days of jardiance changes serum and urinary advanced glycation end product levels
  Other Names: Jardiance
  Arms: Linagliptin
Drug: linagliptin — Test to see how 30 days of tradjenta changes serum and urinary advanced glycation end product levels
  Other Names: tradjenta
  Arms: Empagliflozin

SUMMARY:
Single-center open-label multiple dose randomized two period cross-over study to examine Advanced Glycation End Product (AGE) levels in human subjects pre and post empagliflozin administration.

DETAILED DESCRIPTION:
Single-center open-label multiple dose randomized two period cross-over study.

The North-Shore Long Island Jewish Institutional Review Board will be used to approve our study protocol.

All patients will give written informed consent and comply with the Helsinki agreement and good clinical practices guidelines.

Treatment Plan:

Eligible patients will be randomized to receive linagliptin 5mg daily or empagliflozin 25mg daily for 30 days followed by a 30 day washout period and crossover. All pre-existing diabetic medications will continue unchanged.

Fasting blood carboxymethyl lysine (CML), methylglyoxal (MG), vascular cell adhesion molecule (VCAM), tumor necrosis factor (TNF) alpha, 8-isoprostane, and routine chemistries and urinary CML, MG, and creatinine will be measured at baseline, after 30 days, 60 days and 90 days.

AGE levels will be measured by Elisa.

ELIGIBILITY:
Inclusion Criteria:

* T2DM
* Age ≥ 18
* glomerular filtration rate ≥ 30 ml/min/1.73 m2 body-surface area
* A1C ≥ 7% any higher limit
* SLGT-2 inhibitor naïve
* On stable doses of current medications for at least 3 months.

Exclusion Criteria:

* Indication of liver disease, defined by serum levels of alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase above 2 x upper limit of normal during screening or run-in phase
* Blood dyscrasias or any disorders causing hemolysis or unstable red blood cells
* Contraindications to background therapy according to the local label
* Any uncontrolled endocrine disorder except type 2 diabetes
* Pre-menopausal women (last menstruation ≤1 year prior to informed consent) who were nursing, pregnant, or of child-bearing potential and were not practicing an acceptable method of birth control, or did not plan to continue using this method throughout the study, or did not agree to submit to periodic pregnancy testing during the trial

  o Acceptable methods of birth control include tubal ligation, transdermal patch, intrauterine devices/systems, oral, implantable or injectable contraceptives, sexual abstinence, double barrier method, vasectomy of partner
* Alcohol or drug abuse within 3 months of informed consent that would interfere with trial participation or any ongoing condition leading to decreased compliance with study procedures or study drug intake
* Intake of an investigational drug in another trial within 30 days prior to intake of study medication in this trial or participating in another trial involving an investigational drug and/or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in AGE levels | 30 days
  Measurement of serum and urinary AGE levels

SECONDARY OUTCOMES:
Change in blood pressure | 30 days
  measurement of BP
Change in weight | 30 days
  measurement of weight

IPD SHARING:
Plan to Share IPD: No